CLINICAL TRIAL: NCT02717286
Title: Survival of Restorative Treatment in First Molars Affected by Molar-Incisor Hypomineralization
Brief Title: Restorative Treatment in First Molars Affected by Molar-Incisor Hypomineralization
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal do Paraná (Other)
Responsible Party: Principal Investigator, Juliana Feltrin de Souza Caparroz, Juliana Feltrin de Souza, Universidade Federal do Paraná
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UFParana
Record Dates: First submitted 2016-03-18; First posted 2016-03-23 (Estimated); Last update posted 2016-03-30 (Estimated); Status verified 2016-03

CONDITIONS: Molar Incisor Hypomineralization
MeSH Terms: conditions — Molar Hypomineralization

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (Sham Comparator): 20 first permanent molars from children aged between 6 to 12 years old presenting MIH will be included. A calibrated pediatric dentist examined the selected teeth to classify MIH according to the European Academy of Pediatric Dentistry (EADP) criteria.
  Intervention of Control: The restorative treatment using a total-etching adhesive system, which was performed according to the following operative sequence: prophylaxis, infiltrative anesthesia, rubber dam, application of 37.5% phosphoric acid to enamel (30 s) and dentine (15 s), extensive washing, drying with cotton and air jet (5 s), priming (5 s), light curing (20 s), restoration with composite resin (Filtek XT350), examination of occlusal contact, and final polishing.
  Interventions: Procedure: restorative
- Test (Experimental): 20 first permanent molars from children aged between 6 to 12 years old presenting Molar Incisor Hypomineralization will be included. A calibrated pediatric dentist examined the selected teeth to classify MIH according to the EAPD criteria.
  Intervention of test: the restorative treatment using a self-etching adhesive system, which was performed according to the following operative sequence: prophylaxis, infiltrative anesthesia, rubber dam, application of 37.5% phosphoric acid to enamel (30 s) and dentine (15 s), extensive washing, drying with cotton and air jet (5 s), priming (5 s), air jet (5 s), adhesive application (5 s), light curing (20 s), restoration with composite resin (Filtek XT350), examination of occlusal contact, and final polishing.
  Interventions: Procedure: restorative

INTERVENTIONS:
Procedure: restorative — It was performed direct restoration using two kinds of adhesive system (total-etching adhesive and self-etching adhesive)

SUMMARY:
The restorative management of molars with Molar-Incisor Hypomineralization (MIH) represents a challenge in the clinical practice with high failure rate. Thus, this clinical trial aimed to evaluate the clinical survival of direct composite resin restorations in first permanent molars (FPMs) that are affected by MIH, comparing two adhesive systems.

DETAILED DESCRIPTION:
For the research, it was selected first permanent molars (FPMs) with MIH from children aged 6-8 years. FPM fully erupted and with restorative treatment needed was the inclusion criteria. We excluded FPMs with destroyed crowns. The FPMs were randomly assigned to two groups: G1 (self-etching adhesive) and G2 (total-etching adhesive). Clinical evaluation was performed during 18 months according to the USPHS-Modified by a blinded examiner. The actuarial method was used to evaluate survival of the restorations and Fisher's exact test was used to compare differences between the groups (α=5%).

ELIGIBILITY:
Inclusion Criteria:

* children and/or parents who agree in participate of the study
* children were born and living in Araraquara, SP, Brazil
* presence of the first permanent molars totally erupted with defects classified as enamel post eruptive breakdown (PEB) or unsatisfactory atypical restoration (UATR), with or without carious lesions.

Exclusion Criteria:

* children and/or parents who do not agree in participate of the study
* first permanent molars with enamel malformation associated with syndromes,
* dental fluorosis,
* first permanent molars with destroyed crowns,
* imperfect amelogenesis
* fixed orthodontic appliances.

Ages: 6 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 26 (Actual)
Dates: Start 2013-01; Primary Completion 2013-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Survival rates of the direct restorative treatment | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Rita de Cássia Loiola Cordeiro, PhD, Study Chair — UNESP- Univ Estadual Paulista
Locations (1):
- UNESP - Univ. Estadual Paulista, Araraquara, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes